CLINICAL TRIAL: NCT06444438
Title: Radiological Changes of Glymphatic-meningeal Lymphatic Drainage System After Spontaneous Subarachnoid Hemorrhage
Brief Title: Radiological Changes of Glymphatic-meningeal Lymphatic Drainage System After Subarachnoid Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0224
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-03

CONDITIONS: Subarachnoid Hemorrhage; Lymphatic System Disorder; Meningeal Lymphatic Vessels
MeSH Terms: conditions — Subarachnoid Hemorrhage; Lymphatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ruptured aneurysm: Patients with aneurysmal subarachnoid hemorrhage
  Interventions: Diagnostic Test: subarachnoid hemorrhage
- Unruptured aneurysm: Patients with unruptured aneurysm

INTERVENTIONS:
Diagnostic Test: subarachnoid hemorrhage — CT presented subarachnoid hemorrhage
  Groups: Ruptured aneurysm

SUMMARY:
Subarachnoid hemorrhage (SAH) is a common and extremely critical disease in neurosurgery. The mortality rate within 30 days of the onset of SAH is as high as 50%, and about 15% of SAH patients die without reaching the hospital. Nearly half of the survivors have severe neurological dysfunction, causing a huge burden to the families and society of the patients.

Recently, the introduction of the "glymphatic-meningeal lymphatic vessels" drainage system has updated the current concept of intracranial cerebrospinal fluid circulation. After subarachnoid hemorrhage, a large number of blood components flooded into the subarachnoid space and entered the cerebrospinal fluid circulation, which directly affected the function of the lymphatic-meningeal lymphatic drainage system. Many preclinical animal studies have pointed out that the damage of the lymphatic-meningeal lymphatic drainage system is involved in the aggravation of cerebral edema, neuroinflammation and hydrocephalus after SAH, which ultimately leads to poor prognosis of patients.

However, at present, the changes of the glymphatic-meningeal lymphatic drainage system after SAH have only been confirmed in animal models, and clinical evidence is lacking. With the development of imaging technology, many research teams have confirmed the functional changes of the lymphatic-meningeal lymphatic drainage system in Alzheimer's disease and Parkinson's disease by using different sequences of non-invasive MRI, such as 3D T2-FLAIR, DTI-ALPS and other sequences.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is a common and extremely critical disease in neurosurgery. The mortality rate within 30 days of the onset of SAH is as high as 50% and about 15% of SAH patients die without reaching the hospital. Nearly half of the survivors have severe neurological dysfunction, causing a huge burden to the families and society of the patients.

Recently, the introduction of the "glymphatic-meningeal lymphatic vessels" drainage system has updated the current concept of intracranial cerebrospinal fluid circulation. After subarachnoid hemorrhage, a large number of blood components flooded into the subarachnoid space and entered the cerebrospinal fluid circulation, which directly affected the function of the lymphatic-meningeal lymphatic drainage system. Many preclinical animal studies have pointed out that the damage of the lymphatic-meningeal lymphatic drainage system is involved in the aggravation of cerebral edema, neuroinflammation, and hydrocephalus after SAH, which ultimately leads to poor prognosis of patients.

However, at present, the changes in the glymphatic-meningeal lymphatic drainage system after SAH have only been confirmed in animal models, and clinical evidence is lacking. With the development of imaging technology, many research teams have confirmed the functional changes of the lymphatic-meningeal lymphatic drainage system in Alzheimer's disease and Parkinson's disease by using different sequences of non-invasive MRI, such as 3D T2-FLAIR, DTI-ALPS, and other sequences.

ELIGIBILITY:
Inclusion Criteria:

* ①18-80 years old; ② Voluntary patients with spontaneous subarachnoid hemorrhage undergoing aneurysm interventional therapy.

Exclusion Criteria:

* ①A history of trauma or prior brain injury (stroke, cerebral hemorrhage, etc., leaving associated chronic changes on CT); ②Patients with imaging data loss and severe comorbidities prior to the onset of SAH

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient had no prior brain disease and had a subarachnoid hemorrhage due to a ruptured aneurysm.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The drainage function of the glymphatic system - meningeal lymphatic vessels | Within 7 days after admission
  The drainage function of the lgymphatic system - meningeal lymphatic vessels was observed by magnetic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China